CLINICAL TRIAL: NCT05414188
Title: The Improvement of the Quality of Life and Exercise Capacity Through Pulmonary Rehabilitation in Lung Cancer Patients Receiving Radiation Therapy
Brief Title: Beneficial Effect of Pulmonary Rehabilitation in Lung Cancer Patients Receiving Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Assistant Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0483
Record Dates: First submitted 2022-05-30; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Lung Neoplasm Malignant
Keywords: Pulmonary rehabilitation; Radiation therapy; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation group (Active Comparator): Patients will receive the radiation therapy according to the existing schedule. Additionally, patients in pulmonary rehabilitation group will participate pulmonary rehabilitation program more than two times per week.
  Interventions: Behavioral: Pulmonary rehabilitation
- Control group (No Intervention): Patients will receive the radiation therapy according to the existing schedule. There will be no additional treatment

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — Pulmonary rehabilitation runs for 60 minutes per session. The pulmonary rehabilitation program is based on a comprehensive approach, not simply providing regular exercise. And it includes patient education, active encouragement, and psychological support by investigators. Exercise is performed more than twice a week. Each session is performed for 60 minutes and includes breathing exercises, low to medium-intensity aerobic exercises, and muscle exercises under the guidance of a investigator. After radiation therapy is completed, investigators will recommend that patients perform pulmonary rehabilitation at home more than twice a week and for 60 minutes or more. The patients will record whether and when exercise is performed every day in the diary for pulmonary rehabilitation.
  Arms: Pulmonary rehabilitation group

SUMMARY:
It is important for clinicians to maintain and support for exercise capacity and quality of life of lung cancer patients after radiation therapy, because radiation therapy also affect the lung function and general conditions of patients. The effect and safety of pulmonary rehabilitation is well-proven in various diseases. Because there is no standard treatment, the investigators will perform this study to clearly prove the effect of pulmonary rehabilitation in lung cancer patients receiving radiation therapy.

DETAILED DESCRIPTION:
Roles of the radiation therapy in lung cancer are as followings; 1) to treat the lung caner stage 1 ~2 patients, who are inadequate for operation due to declined lung function, 2) to treat the locally advanced and inoperable stage 3 patients with concurrent chemotherapy, and 3) to palliatively treat the stage 4 patient. However, it is also possible that radiation therapy worsens the general weakness and lung function, although the degree of deterioration was generally less than lung resection. Therefore, it is crucial for clinicians to maintain and support for exercise capacity and quality of life of lung cancer patients after radiation therapy.

The effect and safety of pulmonary rehabilitation is well-proven in various diseases. Investigators presented a retrospective study about the effect of pulmonary rehabilitation in patients receiving radiation therapy, which showed less decreased lung function, less radiation related pneumonitis, and decreased mortality. Investigators will perform this study to clearly prove the effect of pulmonary rehabilitation in lung cancer patients receiving radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Lung cancer patients with scheduled radiation therapy (postoperative adjuvant radiation therapy and concurrent chemoradiation therapy) during more than 4 weeks (5 times a week, 20 times a week)
* Lung parenchymal cancer
* Consent to regular outpatient-based pulmonary rehabilitation program, considering residence and other factors.

Exclusion Criteria:

* Communication restrictions
* Failed to obtain consent form
* Accompanied by psychiatric problems or severe dizziness
* Patients have comorbidities, which are regarded as contraindications of pulmonary rehabilitation, such as severe pulmonary hypertension or hemodynamic instability

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-06-14 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of 6 minutes walking test at 7 months | 7 months
  Change of walking distance from baseline 6 minutes walking test at 7 months

SECONDARY OUTCOMES:
All cause mortality | From the initiation of radiation therapy to 7 months at end of radiation therapy
  All cause mortality during study periods
Radiation therapy related pneumonitis | From the initiation of radiation therapy to 7 months at end of radiation therapy
  Radiation therapy related pneumonitis requiring steroid therapy
Forced Expiratory Volume in 1 sec at 7 months | 7 months
  Forced Expiratory Volume in 1 sec (L, predicted percentage) at 7 months
Forced Expiratory Volume in 1 sec at 1 month | 1 month
  Forced Expiratory Volume in 1 sec (L, predicted percentage) at 1 month
Forced Vital Capacity at 7 months | 7 months
  Forced Vital Capacity (L, predicted percentage) at 7 months
Forced Vital Capacity at 1 month | 1 month
  Forced Vital Capacity (L, predicted percentage) at 1 month
Carbon monoxide diffusing capacity at 7 months | 7 months
  Carbon monoxide diffusing capacity (mL/mmHg/min, predicted percentage) at 7 months
Carbon monoxide diffusing capacity at 1 month | 1 month
  Carbon monoxide diffusing capacity (mL/mmHg/min, predicted percentage) at 1 month
Change of dyspnea scale at 7 months | 7 months
  Investigators will measure the change from the baseline Modified Medical Research Council Dyspnea Scale in the range of 0 to 4, which means the higher the result, the more severe the degree of dyspnea
Change of dyspnea scale at 1 month | 1 month
  Investigators will measure the change from the baseline Modified Medical Research Council Dyspnea Scale in the range of 0 to 4, which means the higher the result, the more severe the degree of dyspnea
Grip strength at 7 months | 7 months
  Grip strength will be measured by digital group hand dynamometer
Grip strength at 1 month | 1 month
  Grip strength will be measured by digital group hand dynamometer
Maximal inspiratory pressure at 7 months | 7 months
  To evaluated respiratory muscle strength, investigators will measure maximal inspiratory pressure by portable spirometry
Maximal expiratory pressure at 7 months | 7 months
  To evaluated respiratory muscle strength, investigators will measure maximal expiratory pressure by portable spirometry
Maximal inspiratory pressure at 1 month | 1 month
  To evaluated respiratory muscle strength, investigators will measure maximal inspiratory pressure by portable spirometry
Maximal expiratory pressure at 1 month | 1 month
  To evaluated respiratory muscle strength, investigators will measure maximal expiratory pressure by portable spirometry
Skeletal muscle mass at 7 months | 7 months
  Investigators will measure the skeletal muscle mass by bioimpedance
Skeletal muscle mass at 1 month | 1 month
  Investigators will measure the skeletal muscle mass by bioimpedance
Appendicular muscle mass at 1 month | 1 month
  Investigators will measure the appendicular muscle mass by bioimpedance
Appendicular muscle mass at 7 months | 7 months
  Investigators will measure the appendicular muscle mass by bioimpedance
Change of The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 at 7 months | 7 months
  Investigators will assess change from the baseline quality of life of patients by questionnaire (The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13) at 7 months. (the higher values indicate a greater degree of symptoms, min.: 0, max.: 100)
Change of The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 at 7 months | 7 months
  Investigators will assess change from the baseline quality of life of patients by questionnaire (The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) at 7 months. (the higher values indicate a greater degree of symptoms, min.: 0, max.: 100)
Change of The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 at 1 month | 1 month
  Investigators will assess change from the baseline quality of life of patients by questionnaire (The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13) at 1 month. (the higher values indicate a greater degree of symptoms, min.: 0, max.: 100)
Change of The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 at 1 month | 1 month
  Investigators will assess change from the baseline quality of life of patients by questionnaire (The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) at 1 month. (the higher values indicate a greater degree of symptoms, min.: 0, max.: 100)
Change of 6 minutes walking test at 1 month | 1 month
  Change of walking distance from baseline 6 minutes walking test at 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jang Ho Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, University of Ulsan College of Medicine, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the primary investigator on reasonable request after end of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Investigators anticipate our study will be finished until December 31, 2023. After end of the study, investigators might consider to share the individual participant data.
Access Criteria: The datasets used and/or analysed during the current study will be available from the primary investigator on reasonable request after end of the study.

REFERENCES:
- [Derived] Lee JH, Cha S, Ko EJ, Kim W, Kim SS, Song SY, Jeon JY, Ji W, Choi CM, Lee SH, Lee SW. Clinical effect of pulmonary rehabilitation during radiotherapy in lung cancer: A randomized controlled trial. Lung Cancer. 2025 Jun;204:108546. doi: 10.1016/j.lungcan.2025.108546. Epub 2025 Apr 17. PMID 40306134